CLINICAL TRIAL: NCT05998434
Title: Home-Based Rehabilitation Training With Human Key-Point Detection for Chronic Low Back Pain Patients: A Randomized Controlled Trial
Brief Title: Home-Based Rehabilitation Training for Chronic Low Back Pain Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Fuming Zheng, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2023]102
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low Back Pain
Keywords: Human Key-Point Detection; Core Stability Exercise; digital healthcare

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the digital therapy (Experimental): The participants randomly assigned to the intervention group will receive home-based exercise training with human key-point detection.They will be instructed to complete a minimum of three sports training sessions per week at their preferred time and location.The exercise prescription will be formulated based on previous comprehensive studies, encompassing exercises targeting strength, balance, flexibility, and mobility.Human key point detection technology accurately estimates 25 key points of the human body in pictures or videos using visual detection.
  Interventions: Behavioral: Improving Low Back Pain Through Motor Control Training
- traditional exercise therapy (Active Comparator): The participants randomly assigned to the control group will receive traditional face-to-face exercise instruction. An experienced therapist( 10 years of experience) will be arranged to provide the subjects with 20-30 minutes of exercise instruction three times a week for four weeks. The training sessions were scheduled to start at 4 p.m. on Monday, Wednesday, and Friday of each week. The exercise training content selected for the control group will be consistent with that of the intervention group.
  Interventions: Behavioral: Improving Low Back Pain Through Motor Control Training

INTERVENTIONS:
Behavioral: Improving Low Back Pain Through Motor Control Training — In the digital healthcare group, participants utilized app-based online motor control training. In contrast, participants in the traditional treatment group underwent motor control training under the guidance of healthcare professionals at the hospital.

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a new digital therapy for managing chronic low back pain in adults. The main questions it aims to answer are:

* Does the digital therapy improve back function and reduce pain intensity in participants with chronic low back pain?
* How does the digital therapy's impact compare to traditional exercise therapy?

Participants in this study will be asked to use the digital therapy app on their smartphones. They will receive guided core stability exercises through the app and will be encouraged to perform these exercises at home. Researchers will assess participants' progress by monitoring their exercise adherence and tracking changes in their back function and pain intensity over time.

To compare the effects of the digital therapy, some participants will follow a traditional exercise therapy program guided by a physical therapist. Researchers will compare the outcomes of these two groups to determine whether the digital therapy is as effective as traditional therapy in improving back function and reducing pain intensity in individuals with chronic low back pain.

DETAILED DESCRIPTION:
This detailed description provides an extended overview of the protocol for the clinical trial focused on testing the efficacy of a digital therapy for managing chronic low back pain. The trial seeks to compare the digital therapy's impact against traditional exercise therapy in individuals with chronic low back pain.

Participants and Procedures:

Participants will be recruited based on specific eligibility criteria, including age, medical history, and duration of chronic low back pain. After obtaining informed consent, participants will be randomly assigned to one of two groups: the digital therapy group or the traditional exercise therapy group.

Digital Therapy Group:

Participants in this group will receive access to a digital therapy app on their smartphones. The app will guide them through core stability exercises, providing step-by-step instructions and visual demonstrations. Participants will be encouraged to perform these exercises regularly at home. Researchers will monitor participants' exercise adherence and collect data on their back function and pain intensity over the study period.

Traditional Exercise Therapy Group:

Participants in this group will receive traditional exercise therapy guided by a physical therapist. They will attend in-person sessions at a designated clinic, where they will receive personalized exercise recommendations and instructions. Similar to the digital therapy group, researchers will monitor exercise adherence and track changes in back function and pain intensity.

Quality Assurance and Data Management:

The study will implement a comprehensive quality assurance plan to ensure the accuracy and reliability of collected data. This plan will include data validation procedures, site monitoring, and auditing. Data checks will be conducted to identify inconsistencies or errors in the collected data. Source data verification will be employed to cross-reference registry data with external sources, such as medical records.

Data Dictionary and Standard Operating Procedures:

A data dictionary will be developed, detailing each variable used in the registry. This will include the source of the variable, coding information, and normal ranges if relevant. Standard Operating Procedures (SOPs) will be established to govern registry operations and analysis activities, covering patient recruitment, data collection, data management, analysis, adverse event reporting, and change management.

Sample Size and Missing Data:

A sample size assessment will be conducted to determine the number of participants or participant years required to demonstrate a statistically significant effect. A plan for handling missing data will be devised to address situations where variables are missing or inconsistent due to various reasons.

Statistical Analysis Plan:

A detailed statistical analysis plan will be developed, outlining the analytical principles and statistical techniques to address primary and secondary objectives outlined in the study protocol or plan. This will guide the analysis of data collected throughout the trial.

In summary, this comprehensive protocol describes the structure, procedures, and quality measures of a clinical trial comparing the effectiveness of a digital therapy and traditional exercise therapy in managing chronic low back pain. The implementation of rigorous quality assurance procedures and data management strategies will ensure the reliability and validity of the study's findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years;
2. Duration of low back pain of at least 12 weeks;
3. Strong willingness to participate in the study and signed informed consent.

Exclusion Criteria:

1. Presence of potential "red flag signs" (e.g., unilateral leg pain and numbness consistent with nerve distribution, intermittent claudication, unexplained sudden weight loss, nocturnal lumbar pain, traumatic lumbago);
2. NRS score less than 4 points;
3. Regular engagement in core stability training in the past four weeks;
4. Inability to independently complete the Chinese electronic questionnaire.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
11-point numeric rating scale（NRS） | baseline，4 weeks and 16 weeks
  NRS;0=no pain, 10=unbearable pain

SECONDARY OUTCOMES:
the Oswestry Disability Index (ODI) | baseline，4 weeks and 16 weeks
  The ODI evaluated disability across 10 domains, encompassing pain intensity and functional abilities related to personal care, lifting, walking, sitting, standing, sleeping, sexual activities, social life, and traveling. Each domain was rated on a 6-point scale ranging from 0 to 5. A score of 0 indicated the highest level of functioning, while a score of 50 indicated total disability
The 36-item Short Form Health Survey (SF-36) | baseline，4 weeks and 16 weeks
  it evaluates an individual's physical, mental, and social health experiences across eight domains, including Physical Functioning, Mental Health, and more. With 36 questions, responses are scored from 0 to 100, reflecting higher scores for better health status. Its brevity, versatility, and comprehensive health dimension coverage are notable advantages. The SF-36 finds applications in clinical practice, epidemiology, and health outcome studies, aiding in diagnosis, treatment, and policy decisions.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuming Z, Zhicheng L, Huanjie H, Xinna Z, Rong C, Jiahui P, Liming Y, Xi C, Chuhuai W. Home-based rehabilitation training with human key point detection for chronic low back pain patients: a randomized controlled trial protocol. Trials. 2023 Nov 27;24(1):760. doi: 10.1186/s13063-023-07805-z. PMID 38012740